CLINICAL TRIAL: NCT03375775
Title: Evaluation of Clinical and Immunological Parameters in Children Treated With Subcutaneous Immunotherapy Towards Pollen - a Controlled Study
Brief Title: Evaluation of Subcutaneous Immunotherapy Towards Pollen in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Maria Ingemansson, Principal Investigator, Karolinska Institutet
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: DNR 2015/3:8 EPN Stockholm
Record Dates: First submitted 2017-11-03; First posted 2017-12-18 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-04

CONDITIONS: Rhinitis, Allergic; Conjunctivitis, Allergic; Asthma
MeSH Terms: conditions — Rhinitis, Allergic; Conjunctivitis, Allergic; Asthma

STUDY DESIGN:
Intervention Model Description: Open controlled study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment group (Experimental): Subcutaneous immunotherapy with ALK Alutard birch or ALK Alutard timothy
  Interventions: Drug: Subcutaneous immunotherapy with ALK Alutard birch or ALK Alutard timothy
- Control group (Active Comparator): No immunotherapy, symptomatic treatment These patients will only receive symptomatic treatment for their allergic rhinoconjunctivitis.
  Interventions: Other: No immunotherapy, symptomatic treatment

INTERVENTIONS:
Drug: Subcutaneous immunotherapy with ALK Alutard birch or ALK Alutard timothy — According to standardized clinical protocol
  Other Names: Subcutaneous immunotherapy with grass and/or birch
  Arms: Treatment group
Other: No immunotherapy, symptomatic treatment — These patients will only receive symptomatic treatment for their allergic rhinoconjunctivitis.
  Arms: Control group

SUMMARY:
The objective is to prospectively explore associations between immunological parameters in blood and clinical effect of subcutaneous immunotherapy (SCIT) in children with severe allergy towards pollen. Half of the children will receive SCIT while the other half will start SCIT after the study is finished. Clinical evaluations of symptoms and an immunological survey will be performed before start of SCIT and after one year of treatment. Some of the immunological parameters will also be checked after 6 months of treatment

DETAILED DESCRIPTION:
Before start of SCIT, with Alutard pollenextract/s from " Allergologisk Laboratorium Köbenhavn" (ALK), and after one year of treatment, immunoglobulin E (IgE)-antibody levels towards the crude allergen and important allergen components in birch and grasspollen (timothy) will be measured in blood. While IgE- antibodies are considered to be an indicator of allergy IgG- and IgG4-antibodies are considered to be "blocking" antibodies in IgE-mediated allergy. Therefore the investigators will measure the IgG- and IgG4-antibody levels to crude allergens and applicable allergen components before start, when maintenance dose is reached (after 6 months) and after one year of treatment. In order to evaluate quality of life, a validated form (DISABKIDS) will be used. Symptom score will be rated by a validated form (LILA). The need for medication to treat allergic rhinitis and asthma will be assessed using questionnaires. A conjunctival provocation with the applicable allergen(s) will be performed before start of SCIT and after one year of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Seasonal Rhinoconjunctivitis caused by grass and/or birch pollen allergy
* Insufficient clinical effect of symptomatic treatment (antihistamine, nasal corticosteroids)
* IgE antibodies to grass and/or birch pollen antigens

Exclusion Criteria:

* severe comorbidity, severe asthma, pregnancy

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Response to a Conjunctival Allergen Challenge | Before treatment and after 12,24 and 36 months
  Change in the dose of allergen needed to elicit a clinical response following ocular administration of the allergen

SECONDARY OUTCOMES:
PADQLQ (pediatric allergic disease quality of life questionnaire) in Swedish LILA | Baseline and after 12,24 and 36 months of immunotherapy
  Includes 26 questions regarding allergic symptoms scored from 0 (no symptoms) to 6 (very severe symptoms) during pollen season. Difference in change of total score between intervention and control group will be assessed
Questionnaire regarding use of pharmacologic treatment for allergy and asthma during pollen season | Baseline and after 12,24 and 36 months of immunotherapy
  Frequency of use of 8 different drugs will be scored from 0(never) to 5 (daily). Difference in change of total score between intervention and control group will be assessed
Questionnaire regarding quality of life | Baseline and after 12,24 and 36 months of immunotherapy
  DISABKIDS, a european quality of life questionnaire used in children with chronic diseases consisting of 37 quality of life questions with answers rated from ever (0=best) to never (5= worst). Difference in change of total score between intervention and control group will be assessed
Change in level of IgE-antibodies | Baseline and after 12,24 and 36 months of immunotherapy
  Difference in change between intervention and control group will be assessed
Change in level of IgG-antibodies | Baseline and after 12,24 and 36 months of immunotherapy
  Difference in change between intervention and control group will be assessed
Change in level of IgG4-antibodies | Baseline and after 12,24 and 36 months of immunotherapy
  Difference in change between intervention and control group will be assessed

CONTACTS AND LOCATIONS:
Overall Officials: Maria Ingemansson, MD, PHD, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Schmid JM, Wurtzen PA, Dahl R, Hoffmann HJ. Pretreatment IgE sensitization patterns determine the molecular profile of the IgG4 response during updosing of subcutaneous immunotherapy with timothy grass pollen extract. J Allergy Clin Immunol. 2016 Feb;137(2):562-70. doi: 10.1016/j.jaci.2015.05.023. Epub 2015 Jun 30. PMID 26141262
- [Result] Borres MP, Ebisawa M, Eigenmann PA. Use of allergen components begins a new era in pediatric allergology. Pediatr Allergy Immunol. 2011 Aug;22(5):454-61. doi: 10.1111/j.1399-3038.2011.01197.x. PMID 21771081
- [Result] Burks AW, Calderon MA, Casale T, Cox L, Demoly P, Jutel M, Nelson H, Akdis CA. Update on allergy immunotherapy: American Academy of Allergy, Asthma & Immunology/European Academy of Allergy and Clinical Immunology/PRACTALL consensus report. J Allergy Clin Immunol. 2013 May;131(5):1288-96.e3. doi: 10.1016/j.jaci.2013.01.049. Epub 2013 Mar 14. PMID 23498595
- [Result] Kiotseridis H, Cilio CM, Bjermer L, Aurivillius M, Jacobsson H, Tunsater A. Swedish translation and validation of the Pediatric Allergic Disease Quality of Life Questionnaire (PADQLQ). Acta Paediatr. 2011 Feb;100(2):242-7. doi: 10.1111/j.1651-2227.2010.02028.x. Epub 2010 Oct 18. PMID 20874810
- [Result] Schmidt S, Debensason D, Muhlan H, Petersen C, Power M, Simeoni MC, Bullinger M; European DISABKIDS Group. The DISABKIDS generic quality of life instrument showed cross-cultural validity. J Clin Epidemiol. 2006 Jun;59(6):587-98. doi: 10.1016/j.jclinepi.2005.09.012. Epub 2006 May 2. PMID 16713521
- [Result] Fauquert JL, Jedrzejczak-Czechowicz M, Rondon C, Calder V, Silva D, Kvenshagen BK, Callebaut I, Allegri P, Santos N, Doan S, Perez Formigo D, Chiambaretta F, Delgado L, Leonardi A; Interest Group on Ocular Allergy (IGOA) from the European Academy of Allergy and Clinical Immunology. Conjunctival allergen provocation test : guidelines for daily practice. Allergy. 2017 Jan;72(1):43-54. doi: 10.1111/all.12986. Epub 2016 Aug 18. PMID 27430124